CLINICAL TRIAL: NCT04648787
Title: A Randomized Intervention Study of Family-integrated Care for Reducing Uncertainty About Illness in Parents of Preterm Infants
Brief Title: A Study of Family-integrated Care for Reducing Uncertainty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: gepingqian
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: traditional nursing with family-integrated care (Experimental): traditional nursing with family-integrated care
  Interventions: Behavioral: family-integrated care
- Control group: traditional nursing (Experimental): traditional nursing
  Interventions: Behavioral: traditional nursing

INTERVENTIONS:
Behavioral: family-integrated care — One week after admission, the parents of premature infants were informed by telephone one day in advance to enter the ward for family participation nursing, and the guidance of daily life nursing for premature infants was given on the same day, including hand hygiene, breast feeding, pacification, changing diapers, bathing and establishment of parent-child relationship. Before discharge, theparents of premature infants should be informed by telephone one day in advance to enter the ward again for family participation nursing, and half a day's guidance was given, including observation and treatment of common symptoms and signs, guidance of home safety prevention and learning to write diary of premature infants.
  Arms: Intervention group: traditional nursing with family-integrated care
Behavioral: traditional nursing — In hospital education: the health education manual for premature infants will be issued at the time of discharge; the patient's condition will be answered by telephone from 14:00 to 16:00 every day.
  Arms: Control group: traditional nursing

SUMMARY:
To explore the intervention effect of family participatory nursing on the uncertainty of illness of parents of hospitalized premature infants, and to evaluate the uncertainty level of parents of premature infants in different stages. The study will be described the feeling of parents of premature infants after family participation nursing through interview. We will provide support for families of premature infants, and then to provide support for growth and development of premature infants.

DETAILED DESCRIPTION:
Most of the current management mode of restricting or forbidding visiting in neonatology, parents can not establish the perception of premature infants and lack of communication with medical staff, which will lead to negative emotions represented by uncertainty of disease.The research on uncertainty of disease started late in China, mostly used in tumor, epilepsy and congenital heart disease. The research on parents of NICU children mostly focused on the analysis of influencing factors of uncertainty of disease, lacking intervention research, and the measures were only the information support mode based on health education. We want to explore the intervention effect of family participatory nursing on the uncertainty of illness of parents of hospitalized premature infants, and to evaluate the uncertainty level of parents of premature infants in different stages. Describe the feeling of parents of premature infants after family participation nursing through interview. We will provide support for families of premature infants, and then to provide support for growth and development of premature infants.

ELIGIBILITY:
Inclusion Criteria:

Children:

* 32 weeks < gestational age < 37 weeks
* Birth weight ≤ 2500g
* Apgar score > 7
* Transferred to our hospital within 8 hours after birth

Parents:

* Have normal communication ability and understanding ability
* Agreed to participate in this study

Exclusion Criteria:

Children:

-With serious life-threatening diseases, the neonatal critical cases score (discussion draft) was rated as "extremely critical"

Parents:

-There are serious diseases or major negative events in the family (such as traffic accidents, natural disasters, etc.)

Ages: 1 Hour to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The total Scores of PPUS(Parents' Perception of Uncertainty Scale ) | from adminssion to discharge (almostly 14 hospitalization days )
  The scale is one of a series of uncertainty scales developed by Mishel in 1998 under the guidance of uncertainty theory of disease, which is one of the series of uncertainty scales for different groups of people. Its content includes 4 dimensions, 31 items, unclear (13 items), complexity (9 items), lack of information (5 items), and unpredictable (4 items). It includes one score from 4 dimensions adding. The score is much higher, the parents maybe feel more uncertainty.According to the response of the responders, from "completely disagree" to "completely agree", the total score is "31-155". The higher the score is, the stronger the uncertainty of the disease is. When the total score is more than 50% of the highest score, the responders are considered to have higher uncertainty of the disease.

SECONDARY OUTCOMES:
The Scores of Family satisfaction | The 30th day after discharge.
  Likert 5-point method was used to score, that is, 2 = very dissatisfied, 4 = dissatisfied, 6 = average, 8 = satisfied and 10 = very satisfied. The satisfaction level of each question was quantified by scoring.satisfied, satisfied and very satisfied with the score of inpatient satisfaction in the total number of discharged children.

OTHER OUTCOMES:
Readmission rate | The 30th day after discharge.
  the proportion of unplanned readmission in the total number of discharged newborns within 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: ping ge qian, bachelor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China